CLINICAL TRIAL: NCT03205709
Title: Cognitive Training and Neuroplasticity in Mild Cognitive Impairment
Acronym: CogTraining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Duke University (Other); Queens College, The City University of New York (Other)
Responsible Party: Principal Investigator, Davangere P. Devanand, Professor of Clinical Psychiatry and Neurology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7395
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment; Memory Disorders; Memory Impairment; Cognitive Impairment; Cognitive Disorder; Cognitive Decline
Keywords: memory; computerized training; cognition; MRI; mci; memory problems; memory complaints
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group 1 (Active Comparator): Computerized Cognitive Training
  Interventions: Other: Computerized Cognitive Training
- Training Group 2 (Placebo Comparator): Crossword puzzles
  Interventions: Other: Crossword Puzzles

INTERVENTIONS:
Other: Computerized Cognitive Training — Computerized online cognitive training will be used to target specific cognitive abilities and neural networks to potentially improve cognitive functioning through neuroplasticity.
  Arms: Training Group 1
Other: Crossword Puzzles — These are intended to mimic crossword puzzles in newspapers.
  Arms: Training Group 2

SUMMARY:
The purpose of this study is to evaluate if systematic cognitive training can improve cognitive performance in participants (55 and older) with memory loss. This study will evaluate the effects of Computerized Cognitive Training (CCT) for improvement in everyday cognitive and function status, in addition to long-term changes in brain networks over an 18-month period. Although there is no distribution of medication for this study, participants are required to have an at-home computer.

DETAILED DESCRIPTION:
In this clinical trial, investigators will evaluate if systematic cognitive training can improve cognitive performance in participants with memory loss. This study is for those who have demonstrated difficulty with memory. It will evaluate the effects of Computerized Cognitive Training (CCT) for improvement in everyday cognitive and function status, in addition to long-term changes in brain networks over an 18-month period. In this study, participants will be randomly assigned to Training Group 1 or 2; therefore, one will have a 50% chance of being assigned to CCT, and a 50% chance of being assigned to Crossword Puzzle Training (CPT). During the 18- month period, participants will be asked to come to the Memory Disorders Clinic at the New York State Psychiatric Institute (NYSPI) for a screening evaluation, and if eligible, will return for five follow-up visits at Weeks 12, 32, 52, and 78.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 55 to 95 years of age (inclusive) at the time of informed consent.
2. Subjective cognitive complaints, i.e., memory or other cognitive complaints, e.g., naming/language.
3. Meets criteria for cognitive impairment defined as scores > 1 below standardized norms on memory function as identified by the Wechsler Memory Scale (WMS) III Logical Memory immediate or delayed recall score.
4. Folstein Mini Mental State score ≥ 23 out of 30.
5. A family member or other individual who is in contact with the patient and consents to serve as informant during the study; this can be a telephone informant in the case of patients who do not have a live-in informant or close significant other.
6. Access to a home desktop or laptop computer at acceptable internet speed for the study duration.

Exclusion Criteria:

1. Diagnosis of dementia of any type.
2. Current clinical evidence of schizophrenia, schizoaffective disorder, major depression, psychosis, or bipolar I disorder (DSM-IV criteria).
3. Active suicidal ideation or plan.
4. Current or recent (past 6 months) alcohol or substance use disorder (DSM-5 criteria).
5. Clinical stroke with residual neurological deficits. While we will not exclude patients with cerebrovascular disease, we will not include patients who have had a stroke with residual clinical deficits because it is not clear that this type of patient is similar to the MCI (Mild Cognitive Impairment) patient generally, and clear-cut neurological impairment, e.g., hemiplegia/hemiparesis or speech impairment, may compromise the patient's ability to do the CCT or active control procedures and to complete the neuropsychological test battery.
6. Use of medications known to have a negative impact on cognition: benzodiazepines in lorazepam equivalents greater than or equal to 1 mg daily, narcotics, anticholinergics. Other patients receive medications that may be associated with cognitive impairment but are rarely considered the likely etiology, e.g., theophylline, nifedipine, beta blockers; they will not be excluded. Patients receiving other psychotropic medications not expected to have a material impact on cognition, e.g., SSRIs (Selective Serotonin Re-uptake Inhibitors) and SNRIs (Serotonin-norepinephrine re-uptake inhibitors) will be eligible.
7. Presence of any of the following disorders: a) Central Nervous System infection, with cerebrospinal fluid evidence of meningitis, encephalitis, or other infectious process; b) dementia of any type; c) Huntington's disease; d) Multiple sclerosis; e) Parkinson's disease; f) Other neurologic disorders with focal signs, e.g., amyotrophic lateral sclerosis; g) Mental retardation.
8. Acute, severe unstable medical illness. For cancer, acutely ill patients (including those with metastases) will be excluded, but past history of successfully treated cancer will not result in exclusion.
9. Contraindication to MRI scan: pacemaker, metal implants following surgery, any other contraindication to MRI. Eligibility for the MRI scan is a requirement for the study.
10. UPSIT (University of Pennsylvania Smell Identification Test) exclusions: current smoker > 1 pack daily, current upper respiratory infection (retested as soon as the infection clears). UPSIT scores are reduced in schizophrenia, Parkinson's disease and Parkinson's related conditions; these disorders are exclusion criteria for this study. Patients with UPSIT exclusions, e.g., current heavy smoker (less than 3% of older adults in our experience), will not receive the UPSIT but will continue to participate in all other aspects of the study.
11. Patients lacking English-speaking ability as determined by self-report and clinical evaluation.
12. Regular online brain training or regular crossword puzzle user, defined as doing these procedures at a frequency of twice weekly or greater during the year prior to screening. Eligible participants who join the trial are instructed not to do these procedures on their own during the trial, i.e., independent of the study.
13. Participation in another intervention trial for cognitive impairment.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davangere P Devanand, MD, Principal Investigator — Columbia University; Murali Doraiswamy, MD, Principal Investigator — Duke University; Joel Sneed, PhD, Principal Investigator — Queens College
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nwosu A, Qian M, Phillips J, Hellegers CA, Rushia S, Sneed J, Petrella JR, Goldberg TE, Devanand DP, Doraiswamy PM. Computerized Cognitive Training in Mild Cognitive Impairment: Findings in African Americans and Caucasians. J Prev Alzheimers Dis. 2024;11(1):149-154. doi: 10.14283/jpad.2023.80. PMID 38230727
- [Derived] Devanand DP, Goldberg TE, Qian M, Rushia SN, Sneed JR, Andrews HF, Nino I, Phillips J, Pence ST, Linares AR, Hellegers CA, Michael AM, Kerner NA, Petrella JR, Doraiswamy PM. Computerized Games versus Crosswords Training in Mild Cognitive Impairment. NEJM Evid. 2022 Dec;1(12):10.1056/evidoa2200121. doi: 10.1056/evidoa2200121. Epub 2022 Oct 27. PMID 37635843
- [Derived] D'Antonio J, Simon-Pearson L, Goldberg T, Sneed JR, Rushia S, Kerner N, Andrews H, Hellegers C, Tolbert S, Perea E, Petrella J, Doraiswamy PM, Devanand D. Cognitive training and neuroplasticity in mild cognitive impairment (COG-IT): protocol for a two-site, blinded, randomised, controlled treatment trial. BMJ Open. 2019 Aug 30;9(8):e028536. doi: 10.1136/bmjopen-2018-028536. PMID 31471436

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Training Group 1 | Training Group 2
Started | 51 | 56
Completed | 44 | 49
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: 107 participants with MCI
Groups:
- Total: Total of all reporting groups
Arm/Group | Training Group 1 | Training Group 2 | Total
Number analyzed (Participants) | 51 | 56 | 107
Age, Customized [Count of Participants; unit: Participants]
  Age ≤70 yr with early MCI | 10 | 11 | 21
  Age ≤70 yr with late MCI | 12 | 14 | 26
  Age >70 yr with early MCI | 11 | 12 | 23
  Age >70 yr with late MCI | 18 | 19 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 17 | 28 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 50 | 53 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 39 | 42 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
MMSE total score [Mean (Standard Deviation); unit: score] — MMSE: Mini Mental State Examination is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30 and the minimum is 0 points. A higher score represents better cognitive function.
  score | 27.1 (1.6) | 26.8 (1.7) | 26.97 (1.6)
ADAS-Cog total score [Mean (Standard Deviation); unit: score] — ADAS-Cog: Alzheimer's Disease Assessment Scale-Cognitive Subscale. The modified ADAS-Cog is a cognitive battery that assesses learning, memory, language production, language comprehension, constructional praxis, ideational praxis, and orientation. Value range: 0-70. A higher score indicates worse cognition.
  score | 9.5 (3.5) | 9.6 (3.5) | 9.6 (3.5)
Neuropsychological composite z-score [Mean (Standard Deviation); unit: units on a scale] — Neuropsychological Testing Composite Score is a composite score of all neuropsychological tests administered in the protocol, i.e. Auditory Verbal Learning Test, Block Design, Verbal Fluency, Visual Reproduction, Boston Naming Task, Trails A and B. As per standard z-score calculations, the z-score has a mean value of 0 and a SD of 1.
  units on a scale | -0.1 (1.0) | 0.1 (1.0) | 0 (1.0)
UPSA total score [Mean (Standard Deviation); unit: score] — UPSA: UCSD Performance-Based Skills Assessment, range 0-100, higher scores indicate better cognitive function. This is a role-play test designed to evaluate a person's functional capacity in the communication and finance areas of basic living skills.
  score | 80.6 (10.9) | 81.5 (11.4) | 81.1 (11.1)
FAQ total score [Mean (Standard Deviation); unit: score] — FAQ: Functional Activities Questionnaire (FAQ) measures instrumental activities of daily living (IADLs), such as preparing balanced meals and managing personal finances. The score ranges from 0-30. A higher score indicates a greater level of impairment in the instrumental activities of daily living.
  score | 3.4 (4.1) | 3.2 (3.9) | 3.26 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog)
Description: The modified ADAS-Cog is a cognitive battery that assesses learning, memory, language production, language comprehension, constructional praxis, ideational praxis, and orientation. Value range: 0-70. A higher score indicates worse cognition.
Time Frame: [Time Frame: 78 weeks]
Population: Participants assessed at baseline and week 78, and the change over 78 weeks is the outcome.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Training Group 1 | Training Group 2
Number analyzed (Participants) | 44 | 51
score | -0.89 (0.51) | 0.55 (0.48)

2. Secondary Outcome: Change Over Time in Neuropsychological Testing Composite Score
Description: Neuropsychological Testing Composite Score is a compiled score of all neuropsychological tests administered in the protocol, i.e. Auditory Verbal Learning Test, Block Design, Verbal Fluency, Visual Reproduction, Boston Naming Task, Trails A and B.
  The composite neuropsychological test battery is derived by computing the baseline z-score for each individual test and then averaging the resulting z scores. The range will be -5 to +5. z score of 0 represents the sample mean and higher z score indicates better performance.
Time Frame: [Time Frame: Week 78]
Population: Participants assessed at baseline and week 78, and the change over 78 weeks is the outcome.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Training Group 1 | Training Group 2
Number analyzed (Participants) | 51 | 56
score | -0.24 (0.08) | -0.27 (0.07)

3. Secondary Outcome: Change Over Time in Functional Activities Questionnaire (FAQ)
Description: FAQ: Functional Activities Questionnaire (FAQ) measures instrumental activities of daily living (IADLs), such as preparing balanced meals and managing personal finances. The score ranges from 0-30. A higher score indicates a greater level of impairment in the instrumental activities of daily living.
Time Frame: [Time Frame: week 78]
Population: Participants assessed at baseline and week 78, and the change over 78 weeks is the outcome.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Training Group 1 | Training Group 2
Number analyzed (Participants) | 51 | 56
score | -2.00 (0.34) | -0.92 (0.31)

4. Secondary Outcome: Change Over Time in UCSD Performance-Based Skills Assessment (UPSA)
Description: UPSA: UCSD Performance-Based Skills Assessment. The UPSA is a performance-based measure of functional abilities that includes measures of simulated real-world activities, for example, planning a trip to the beach, remembering documents to bring to a medical appointment, and dialing a phone number. A higher score indicates greater cognitive function.
  For the UPSA the z score at baseline is computed (based on the mean and SD of the raw scores). The expected range is -5 to +5 with z score of 0 representing the sample mean and higher z score indicating better performance.
Time Frame: [Time Frame: week 78]
Population: Participants assessed at baseline and week 78, and the change over 78 weeks is the outcome.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Training Group 1 | Training Group 2
Number analyzed (Participants) | 51 | 56
score | 0.55 (1.23) | -0.99 (1.44)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant throughout the study participant duration of 78 weeks.
Description: The definitions used to collect adverse event information in this study align with those from the clinicaltrials.gov definitions.
  Adverse events were reported to research staff and study physicians. These adverse events were recorded, reported per the IRB guidelines, and assessed by the study DSMB.
Arm/Group | Training Group 1 | Training Group 2
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/56
Serious Adverse Events (participants affected / at risk) | 12/51 | 9/56
Other Adverse Events (participants affected / at risk) | 19/51 | 23/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Training Group 1 (N=51) | Training Group 2 (N=56)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (1)
Falls (General disorders) | 2 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac disorders (Cardiac disorders) | 0 (0) | 2 (2)
Vascular disorders (Vascular disorders) | 3 (3) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary disorder (Renal and urinary disorders) | 0 (0) | 2 (2)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Training Group 1 (N=51) | Training Group 2 (N=56)
Fatigue (General disorders) | 2 (3) | 2 (2)
Falls (General disorders) | 2 (4) | 1 (1)
Eye disorders (Eye disorders) | 1 (1) | 4 (5)
Ear, nose, throat disorders (Ear and labyrinth disorders) | 2 (3) | 2 (2)
Skin cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hematological/immune disorders (Immune system disorders) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Elective cardiac surgery (Cardiac disorders) | 1 (1) | 2 (3)
Urinary tract disorders (Renal and urinary disorders) | 0 (0) | 2 (4)
Arthritis, musculoskeletal symptoms (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 2 (3) | 2 (2)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
COVID-19 diagnosis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03205709/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT03205709/SAP_001.pdf
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03205709/ICF_002.pdf